CLINICAL TRIAL: NCT07077889
Title: Incidence and Risk Factors of Chronic Postoperative Pain in Gynaecological Cancer Surgery: a Retrospective Study
Brief Title: Postoperative Chronic Pain in Gynaecological Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Duygu Akyol (Other Government)
Responsible Party: Sponsor-Investigator, Duygu Akyol, Principal investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Organization: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Other Study IDs: 2025-221
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2024-01

CONDITIONS: Gynecologic Cancers; Postoperative Pain
Keywords: gynecological cancer surgery; chronic postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing gynecologic cancer surgery: postoperative chronic pain in patients operated for gynaecological cancer

SUMMARY:
The aim of this study was to determine the incidence of postoperative chronic pain in gynaecological cancer surgery and the analgesia methods used for postoperative analgesia.

The main question(s) aimed to be answered are:

[Which analgesia method has the lowest incidence of postoperative chronic pain?] Patients undergoing gynaecological cancer surgery were retrospectively reviewed. The investigators evaluated the analgesia methods used for postoperative analgesia and the incidence of postoperative chronic pain.

DETAILED DESCRIPTION:
This study was designed retrospectively. The investigators evaluated analgesia methods in patients undergoing surgery for gynaecological cancer between January 2024 and July 2025. In this study, the investigators planned to evaluate the incidence of postoperative chronic pain by evaluating patients for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Gynaecological cancer surgery
* >18 years

Exclusion Criteria:

* Incomplete or inadequate patient records

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The incidence of postoperative chronic pain after surgery was evaluated in patients operated for gynaecological cancer between January 2024 and December 2025.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-07-12 (Actual); Study Completion 2025-07-12 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative chronic pain | 3 months postoperatively
  In our study, the investigators aimed to evaluate the incidence of postoperative chronic pain in patients operated for gynaecological cancer. for this purpose, postoperative patients were contacted at the end of 3 months and the presence of pain was evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: DUYGU AKYOL, M.D, Principal Investigator — Başakşehir Çam & Sakura City Hospital
Locations (1):
- Basaksehir Cam and Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ladjevic N, Milinic M, Jovanovic V, Jovicic J, Likic I, Ladjevic N. CHRONIC POSTOPERATIVE PAIN. Acta Clin Croat. 2023 Nov;62(Suppl4):88-96. doi: 10.20471/acc.2023.62.s4.13. PMID 40463450
- [Background] Gomez M, Izquierdo CE, Mayoral Rojals V, Pergolizzi J Jr, Plancarte Sanchez R, Paladini A, Varrassi G. Considerations for Better Management of Postoperative Pain in Light of Chronic Postoperative Pain: A Narrative Review. Cureus. 2022 Apr 2;14(4):e23763. doi: 10.7759/cureus.23763. eCollection 2022 Apr. PMID 35518528
- [Background] Lopes A, Seligman Menezes M, Antonio Moreira de Barros G. Chronic postoperative pain: ubiquitous and scarcely appraised: narrative review. Braz J Anesthesiol. 2021 Nov-Dec;71(6):649-655. doi: 10.1016/j.bjane.2020.10.014. Epub 2021 Feb 18. PMID 34715995
- [Background] Treede RD, Rief W, Barke A, Aziz Q, Bennett MI, Benoliel R, Cohen M, Evers S, Finnerup NB, First MB, Giamberardino MA, Kaasa S, Korwisi B, Kosek E, Lavand'homme P, Nicholas M, Perrot S, Scholz J, Schug S, Smith BH, Svensson P, Vlaeyen JWS, Wang SJ. Chronic pain as a symptom or a disease: the IASP Classification of Chronic Pain for the International Classification of Diseases (ICD-11). Pain. 2019 Jan;160(1):19-27. doi: 10.1097/j.pain.0000000000001384. PMID 30586067